CLINICAL TRIAL: NCT06741657
Title: A Randomized, Open-Label, 2-Arm, 2-Part, Parallel Group Study to Assess the Pharmacokinetic Comparability of Subcutaneously Administered Litifilimab (BIIB059) Delivered by 3 Devices (Pre-Filled Syringe, Autoinjector, or On-Body Injector) in Healthy Participants
Brief Title: A Study to Find Out How Litifilimab is Processed in the Body in Healthy Participants When Given Under the Skin in 3 Different Ways
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 230HV102
Record Dates: First submitted 2024-12-15; First posted 2024-12-19 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: AI versus PFS (Experimental): Participants will receive SC dose of litifilimab injection via AI or PFS on Day 1 of the study.
  Interventions: Drug: Litifilimab; Device: AI; Device: PFS
- Part 2: OBI versus PFS (Experimental): Participants will receive SC dose of litifilimab injection via OBI or PFS on Day 1 of the study.
  Interventions: Drug: Litifilimab; Device: OBI; Device: PFS

INTERVENTIONS:
Drug: Litifilimab — Administered as specified in the treatment arm.
  Other Names: BIIB059
Device: AI — Administered as specified in the treatment arm.
  Arms: Part 1: AI versus PFS
Device: OBI — Administered as specified in the treatment arm.
  Arms: Part 2: OBI versus PFS
Device: PFS — Administered as specified in the treatment arm.

SUMMARY:
In this study, researchers will learn how the body processes litifilimab when it is given under the skin in 3 different ways. Currently, ongoing studies utilize pre-filled syringes (PFS) that can deliver litifilimab subcutaneously (SC), also known as under the skin.

In this study, researchers want to learn more about new ways of delivering litifilimab SC using either an autoinjector (AI) or an on-body injector (OBI):

Both devices are designed to deliver litifilimab in an automatic way, especially helping patients who may not be able to use their hands very well, or who may be afraid of needles. While the AI is handheld, the OBI device works by being placed on the skin and can help deliver the highest amount of litifilimab through a single injection. The main objective of this study is to learn how the body processes litifilimab after using the AI device or the OBI device, as compared to using the PFS method.

The main questions researchers want to answer are:

* What is the highest amount of litifilimab found in the blood after dosing? How much total litifilimab is found in the blood throughout the study? Researchers will also learn more about: Any medical problems the participants have during the study
* Any injection site pain or reactions the participants may have. Any skin reactions to the OBI device
* Any changes in the participants' overall health after receiving litifilimab.

This study will be done as follows:

* Participants will be screened to check if they can join the study. The screening period will be up to 4 weeks, after which selected participants will check into their study research center.
* Participants will be randomly assigned to be in Part 1 or Part 2 of the study:
* Part 1: Participants will receive SC injection(s) of litifilimab through either the AI device or through PFS.
* Part 2: Participants will receive SC injection(s) of litifilimab through the OBI device or through PFS.
* Participants will remain at their study research center for the first 8 days. After that, there will be a follow-up period for 17 weeks during which participants return to the center a total of 6 times.

Each participant will be in the study for about 22 weeks.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the pharmacokinetic (PK) comparability of litifilimab administered via SC injection(s) of AI (Test Device 1) or SC injection(s) of OBI (Test Device 2), with SC injections of PFS (Reference) in healthy participants.

The secondary objectives of this study are to evaluate the safety and tolerability following SC dose of litifilimab via AI, OBI, or PFS; to assess additional PK parameters following SC dose of litifilimab via AI, OBI, or PFS in healthy participants.

ELIGIBILITY:
Key Inclusion Criteria

* Must have a body mass index between 18.5 and 30 kilograms per square meter (kg/m^2), and a body weight ≥ 50 kg to ≤ 100 kg.
* Must be in good health as determined by the investigator, based on medical history physical examination, electrocardiogram (ECG), and other screening evaluations.

Key Exclusion Criteria

* History of any clinically significant cardiac, endocrine, gastrointestinal, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, or renal disease, or other major disease, as determined by the investigator.
* A positive diagnostic tuberculosis test result within 4 weeks prior to Enrollment (Day 1), defined as a positive QuantiFERON® test result or 2 successive indeterminate QuantiFERON test results.
* History or positive test result for human immunodeficiency virus (HIV).
* History of severe herpes infection such as herpetic encephalitis, ophthalmic herpes, or disseminated herpes.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 404 (Actual)
Dates: Start 2025-01-02 (Actual); Primary Completion 2026-04-08 (Estimated); Study Completion 2026-04-08 (Estimated)

PRIMARY OUTCOMES:
Part 1 and 2: Maximum Observed Concentration (Cmax) of Litifilimab | Pre-dose and at multiple timepoints up to Week 22
Part 1 and 2: Area Under the Concentration-Time Curve From Time 0 to Infinity (AUC0-inf) | Pre-dose and at multiple timepoints up to Week 22

SECONDARY OUTCOMES:
Part 1 and 2: Number of Participants with Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | From screening up to Week 22
Part 1 and 2: Change From Baseline in the Injection Site Pain as Measured by Patient Reported Outcome (PRO) Using a Pain Intensity Numeric Rating Scale (PI-NRS) | Baseline, Day 1
  A PI-NRS scale will be used to assess overall injection site pain at different time points. The scale ranges from 0 to 10 where '0' indicates 'no pain' and '7-10' indicates 'severe pain'.
Part 1 and 2: Percentage of Participants With Mild, Moderate, Severe, or no Injection Site Reactions | Up to Week 1
Part 2: Percentage of Participants With Adhesive Contact Skin Reactions as Measured by Dermal Response and Other Effects Scales | Up to Week 1
  A dermal response scale will be used to assess the adhesive contact skin reactions. The scale ranges from 0 to 7, where '0' indicates 'no evidence of irritation' and '7' indicates 'strong reaction spreading beyond the application site'. The other effects scale ranges from 'A(0)' to 'H(3)', where a 'A(0)' indicates a slightly glazed appearance and 'H(3)' indicates small petechial erosions and/or scabs.
Part 1 and 2: Number of Participants With Change From Baseline in Clinically Significant Vital Signs Abnormalities | Baseline, up to Week 22
Part 1 and 2: Number of Participants With Change From Baseline in Clinically Significant 12-Lead Electrocardiograms (ECGs) Abnormalities | Baseline, up to Week 4
Part 1 and 2: Number of Participants With Change From Baseline in Clinically Significant Laboratory Evaluation Abnormalities | Baseline, up to Week 22
Part 1 and 2: Number of Participants With Change From Baseline in Clinically Significant Physical Examination Abnormalities | Baseline, up to Week 22
Part 1 and 2: Time to Reach Cmax (Tmax) of Litifilimab | Pre-dose and at multiple timepoints up to Week 22
Part 1 and 2: Terminal Elimination Half-life (t1/2) of Litifilimab | Pre-dose and at multiple timepoints up to Week 22
Part 1 and 2: Apparent Total Clearance (CL/F) of Litifilimab | Pre-dose and at multiple timepoints up to Week 22
Part 1 and 2: Volume of Distribution (Vd/F) of Litifilimab | Pre-dose and at multiple timepoints up to Week 22
Part 1 and 2: Area Under the Concentration-Time Curve From Time 0 to the Last Measurable Concentration (AUC0-last) of Litifilimab | Pre-dose and at multiple timepoints up to Week 22

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (2):
- United States (2):
  - Las Vegas Clinical Research Unit, Las Vegas, Nevada
  - Austin Clinical Research Unit, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/